CLINICAL TRIAL: NCT00226434
Title: Early vs Late Introduction of Antiretroviral Therapy in Naive HIV-infected Patients With Tuberculosis in Cambodia
Brief Title: Early vs Late Introduction of Antiretroviral Therapy in HIV-infected Patients With Tuberculosis (ANRS 1295 CAMELIA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Organization: ANRS, Emerging Infectious Diseases (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 1295 CAMELIA; CIPRA KH 001; NCT00498823 (obsolete NCT alias); NCT01300481 (obsolete NCT alias)
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: HIV Infection; Tuberculosis
Keywords: HIV infection; Tuberculosis; Paradoxical reaction; Treatment Naive
MeSH Terms: conditions — HIV Infections; Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Procedure: Early antiretroviral treatment
- 2 (Active Comparator)
  Interventions: Procedure: Late antiretroviral treatment

INTERVENTIONS:
Procedure: Early antiretroviral treatment — The ARV treatment is started 2 weeks after the diagnosis and the start of the anti-tuberculosis treatment
  Arms: 1
Procedure: Late antiretroviral treatment — The ARV treatment is started 8 weeks after the diagnosis and the start of the anti-tuberculosis treatment
  Arms: 2

SUMMARY:
In Cambodia the prevalence of both tuberculosis (TB) and Human Immunodeficiency Virus (HIV) infection is high. Data suggest that aggressive management of HIV infection, which includes Anti-Retroviral Therapy (HAART) during treatment of TB, decreases both morbidity and mortality. On the other hand, the use of HAART for patients with TB may cause severe complications due to drug-drug interactions, and occasionally a temporary exacerbation of symptoms. These reactions may be particularly severe when HAART is started soon after the start of TB treatment.

The proposed study aims to determine the optimal time to initiate HAART in previously untreated HIV-infected adult patients with TB and low CD4 cell counts.

DETAILED DESCRIPTION:
In Cambodia the prevalence of both tuberculosis (TB) and Human Immunodeficiency Virus (HIV) infection is high. In 2000, there were approximately 75.000 newly diagnosed TB cases. In 2003, 1.9% of the population was infected with HIV. TB rates in Cambodia are more than double those observed in other developing countries and up to 30 times higher than those currently seen in the USA or Western Europe. It is estimated that over 8% of the newly diagnosed TB cases are co-infected with HIV, of which approximately 85% are severely immunosuppressed (CD4+ cell count < 200 x 106 cells/l).

Mortality rates were found to be 2-4 folds higher in HIV/TB co-infected patients than in TB alone. Data suggest that aggressive management of HIV infection, which includes Highly Active Anti-Retroviral Therapy (HAART) during treatment of TB decreases both morbidity and mortality by suppressing viral replication and improving immune function.

On the other hand, the use of HAART for patients with TB may cause severe complications due to drug-drug interactions, and occasionally a temporary exacerbation of symptoms, signs or radiographic manifestations of TB. Such events or 'paradoxical reactions' that occur among 7 - 36% of HIV/TB co-infected patients treated with HAART may be secondary to immune restitution. These reactions may be particularly severe when HAART is started soon after the start of TB treatment.

Most clinical teams recommend delaying the initiation of HAART to avoid the early side effects of TB treatment and simplify clinical management of the co-infected patient. However others argue that early initiation of HAART in TB patients with CD4 cell counts < 100 x 106 cells/l leads to a marked reduction of viral load despite frequent adverse events.

The proposed study aims to determine the optimal time to initiate HAART (defined as d4T + 3TC + efavirenz) in previously untreated HIV-infected adult patients with TB and low CD4 cell counts. The study is a multicentre prospective, randomized, open-label two-armed trial with no placebo. It is designed as a superiority trial to compare the "early arm" (HAART initiated 2 weeks after TB treatment onset) with the "late arm" (HAART initiated 2 months after TB treatment onset). Efficacy will be assessed by the survival rate in the two arms. Secondary objectives will include evaluation of (1) the safety of an early initiation of HAART in terms of drug interactions or paradoxical reactions, (2) the occurrence of opportunistic infections diagnosed during the follow-up period, (3) patients' adherence to TB treatment and HAART, (4) the rate of hospitalization for any cause during the trial; the measure of (5) the effectiveness of the TB treatment and HAART and (6) the predictive factors for the survival, the response to anti-TB therapy and HAART and the paradoxical reactions.

The total study duration is expected to be 4 years (3 years for enrolment and at least one year of follow-up) in five study sites: (1) Khmero-Soviet Friendship Hospital, Phnom Penh; (2) Calmette Hospital, Phnom Penh; (3) Provincial hospital, Svay Rieng province; and (4) Provincial hospital, Takeo province, (5) Provincial Hospital, Siem Reap.

The study will be carried out in compliance with the protocol and in accordance with the Declaration of Helsinki approved by the World Health Association and with the recommendations of the Good Clinical Practice.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* Positive HIV test result
* CD4+ cell count under or equal to 200 cells per ml within 14 days prior the study entry
* Positive AFB on any smear (sputum, lymph node drainage, stool, CSF, pleural fluid)
* Naive to ART
* TB treatment started less than one week prior enrolment
* Negative gonadotrophin pregnancy test (blood) for women of childbearing potential (i.e. not surgically sterile or less than 2 years menopause)
* Agreement from female candidates who are participating in sexual activity that could lead to pregnancy while receiving and for 6 weeks after stopping efavirenz to use two reliable methods of contraception, one of which including condom.

Exclusion Criteria:

* Suspected TB with negative AFB
* Pregnant or breastfeeding women
* Impaired hepatic function (icterus, elevated AST or ALT at least 5 times over the normal value)
* Unable and/or unlikely to comprehend and/or be adherent to the protocol
* Treated for a previous suspected or documented TB other than the ongoing infection which motivates enrolment in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 661 (Actual)
Dates: Start 2006-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Survival rate | At the end of the study

SECONDARY OUTCOMES:
Type, frequency and severity of Adverse Events that occur during the trial and to their potential relations with the drugs, HIV or TB infection | During the overall study
Frequency of Immune Reconstitution Inflammatory Syndrome | During the overall study
Frequency of TB paradoxical reaction, defined as worsening or emergence of signs or symptoms of TB (e.g. fever, cough, shortness of breath, adenopathy or exacerbation of disease at other extra pulmonary sites) during appropriate TB treatment | During the overall study
Occurrence of opportunistic infections | During the overall study
Evaluation of TB treatment success | During the overall study
Evaluation of ART treatment success | During the overall study
Resistance to ARV treatment determined by genotyping HIV-1 strains among patients with detectable viral load on Day 0 and Week 50 | Within 12 months of follow-up
Patient's adherence to TB and ARV treatment evaluated based on interviews and pill counts at each study visit | During the overall study
Pharmacokinetic study to assess efavirenz plasma exposure will be assayed at regular time intervals | Within 12 months of follow-up
Survival Rate | 50 weeks after enrolment

CONTACTS AND LOCATIONS:
Overall Officials: François-Xavier Blanc, Principal Investigator — Bicêtre University Hospital, France; Thim Sok, Principal Investigator — Cambodian Health Committee, Phnom Penh, Cambodia; Anne Goldfeld, Principal Investigator — Institute for Biomedical Research, Boston, USA
Locations (5):
- Cambodia (5):
  - Calmette Hospital, Phnom Penh
  - Khmero-Soviet Friendship Hospital, Phnom Penh
  - Siem Reap Referral Hospital, Siem Reap
  - Provincial hospital, Svay Rieng
  - Provincial hospital, Takeo

REFERENCES:
- [Background] Blanc FX, Havlir DV, Onyebujoh PC, Thim S, Goldfeld AE, Delfraissy JF. Treatment strategies for HIV-infected patients with tuberculosis: ongoing and planned clinical trials. J Infect Dis. 2007 Aug 15;196 Suppl 1:S46-51. doi: 10.1086/518658. PMID 17624825
- [Derived] Marcy O, Laureillard D, Madec Y, Chan S, Mayaud C, Borand L, Prak N, Kim C, Lak KK, Hak C, Dim B, Sok T, Delfraissy JF, Goldfeld AE, Blanc FX; CAMELIA (ANRS 1295-CIPRA KH001) Study Team. Causes and determinants of mortality in HIV-infected adults with tuberculosis: an analysis from the CAMELIA ANRS 1295-CIPRA KH001 randomized trial. Clin Infect Dis. 2014 Aug 1;59(3):435-45. doi: 10.1093/cid/ciu283. Epub 2014 Apr 23. PMID 24759827
- [Derived] Borand L, Madec Y, Laureillard D, Chou M, Marcy O, Pheng P, Prak N, Kim C, Lak KK, Hak C, Dim B, Nerrienet E, Fontanet A, Sok T, Goldfeld AE, Blanc FX, Taburet AM. Plasma concentrations, efficacy and safety of efavirenz in HIV-infected adults treated for tuberculosis in Cambodia (ANRS 1295-CIPRA KH001 CAMELIA trial). PLoS One. 2014 Mar 7;9(3):e90350. doi: 10.1371/journal.pone.0090350. eCollection 2014. PMID 24608960
- [Derived] Laureillard D, Marcy O, Madec Y, Chea S, Chan S, Borand L, Fernandez M, Prak N, Kim C, Dim B, Nerrienet E, Sok T, Delfraissy JF, Goldfeld AE, Blanc FX; CAMELIA (ANRS 1295 - CIPRA KH001) Study Team. Paradoxical tuberculosis-associated immune reconstitution inflammatory syndrome after early initiation of antiretroviral therapy in a randomized clinical trial. AIDS. 2013 Oct 23;27(16):2577-86. doi: 10.1097/01.aids.0000432456.14099.c7. PMID 24096631
- [Derived] Borand L, Laureillard D, Madec Y, Chou M, Pheng P, Marcy O, Sok T, Goldfeld AE, Taburet AM, Blanc FX; CAMELIA ANRS 1295-CIPRA KH001 Study Team. Plasma concentrations of efavirenz with a 600 mg standard dose in Cambodian HIV-infected adults treated for tuberculosis with a body weight above 50 kg. Antivir Ther. 2013;18(3):419-23. doi: 10.3851/IMP2483. Epub 2012 Dec 12. PMID 23237982
- [Derived] Blanc FX, Sok T, Laureillard D, Borand L, Rekacewicz C, Nerrienet E, Madec Y, Marcy O, Chan S, Prak N, Kim C, Lak KK, Hak C, Dim B, Sin CI, Sun S, Guillard B, Sar B, Vong S, Fernandez M, Fox L, Delfraissy JF, Goldfeld AE; CAMELIA (ANRS 1295-CIPRA KH001) Study Team. Earlier versus later start of antiretroviral therapy in HIV-infected adults with tuberculosis. N Engl J Med. 2011 Oct 20;365(16):1471-81. doi: 10.1056/NEJMoa1013911. PMID 22010913